CLINICAL TRIAL: NCT03069456
Title: Comparative Population Pharmacodynamic Modeling for Sevoflurane Effects Using Anesthetic Depth Monitoring for Sedation (ADMS) and Bispectral Index System (BIS)
Brief Title: Comparative Population Pharmacodynamic Modeling for Sevoflurane Effects Using ADMS and Bispectral Index
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Seongwook Jeong, professor, Chonnam National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CNUHH-2015-067
Record Dates: First submitted 2017-02-15; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Anesthesia
Keywords: sevoflurane; Bistpectral index; Anesthetic Depth Monitoring System; population pharmacodynamics

STUDY DESIGN:
Intervention Model Description: Combined sigmoidal Emax models from anesthetic depth monitoring for sedation (ADMS) and combined sigmoidal Emax models from bispectral index (BIS) via population pharmacodynamic approach.
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIS group (Active Comparator): Combined sigmoidal Emax models from the BIS data
  Interventions: Device: BIS
- ADMS group (Experimental): Combined sigmoidal Emax models from the ADMS data
  Interventions: Device: ADMS

INTERVENTIONS:
Device: BIS
  Arms: BIS group
Device: ADMS
  Arms: ADMS group

SUMMARY:
The investigators want to compare the performance of anesthetic depth monitoring for sedation (ADMS) to the bispectral index (BIS) as electroencephalographic measures of sevoflurane effect using two combined sigmoidal Emax models via population pharmacodynamic approach.

DETAILED DESCRIPTION:
Intraoperative awareness under general anesthesia is rare, but it may cause serious psychological sequelae. Anesthetic depth monitoring system based on electroencephalography(EEG) or evoked potential are broadly used methods. Bispectral index (BIS) monitor is most popular anesthetic depth monitoring system. Anesthetic depth monitoring for sedation (ADMS) is developed in Korea as an electroencephalographic monitor for measuring the depth of anesthesia. The investigators want to compare the performance of ADMS to the bispectral index (BIS) as electroencephalographic measures of sevoflurane effect using two combined sigmoidal Emax models via population pharmacodynamic approach.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for an elective operation and postoperative epidural PCA with ASA physical status 1,2,3 who have signed the wrtten informed consent.

Exclusion Criteria:

* preventive anticoagulation treatment
* Significant liver, kidney, coagulation dysfunction
* Clinically significant ECG abnormalities
* administration of psychologic durgs or opioid within 14 days before surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Bispectral Index (BIS) | Data capture will be started 45 minutes after induction of general anesthesia for 70 minutes
  captured BIS data (0~100) from the BIS system after induction of general anesthesia, sevoflurane concentrations will be progressively increased and then decreased over 70 min.
Anesthetic depth monitoring for sedation (ADMS) | Data capture will be started 45 minutes after induction of general anesthesia for 70 minutes
  captured ADMS data (0~100) from the ADMS system after induction of general anesthesia, sevoflurane concentrations will be progressively increased and then decreased over 70 min.

SECONDARY OUTCOMES:
Adverse events | visit patients 24 hours after operation.
  Observe all adverse events both groups

CONTACTS AND LOCATIONS:
Overall Officials: SEONGWOOK JEONG, MD, PhD., Principal Investigator — Chonnam National University Hospital
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han DW, Linares-Perdomo OJ, Lee JS, Kim JH, Kern SE. Comparison between cerebral state index and bispectral index as measures of electroencephalographic effects of sevoflurane using combined sigmoidal E(max) model. Acta Pharmacol Sin. 2011 Oct;32(10):1208-14. doi: 10.1038/aps.2011.99. Epub 2011 Sep 5. PMID 21892201
- [Background] Kreuer S, Bruhn J, Wilhelm W, Grundmann U, Rensing H, Ziegeler S. Comparative pharmacodynamic modeling of desflurane, sevoflurane and isoflurane. J Clin Monit Comput. 2009 Oct;23(5):299-305. doi: 10.1007/s10877-009-9196-6. Epub 2009 Aug 27. PMID 19711188
- [Background] Rehberg B, Bouillon T, Zinserling J, Hoeft A. Comparative pharmacodynamic modeling of the electroencephalography-slowing effect of isoflurane, sevoflurane, and desflurane. Anesthesiology. 1999 Aug;91(2):397-405. doi: 10.1097/00000542-199908000-00013. PMID 10443602